CLINICAL TRIAL: NCT03207711
Title: Optimizing Lifestyle Interventions With Mindfulness-based Strategies in Type 2 Diabetes
Brief Title: Delish Study: Diabetes Education to Lower Insulin, Sugars, and Hunger
Acronym: Delish
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R61AT009333 (NIH); R61AT009333 (NIH)
Record Dates: First submitted 2017-06-11; First posted 2017-07-05 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet, Carbohydrate-Restricted; Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blood tests at LabCorp and 24-hour dietary recall interviews are done by research assistants blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet Education (Active Comparator): All participants will receive instruction in the carbohydrate-restricted diet (CR).The study diet has approximately 10% of kcal coming from carbohydrate, typically 50 grams/day or fewer, not including fiber. Participants will be encouraged to eat a normal amount of protein, typically about 80-100 grams/day (about 20-25% of calories), and the rest of their calories from fat. Foods that are encouraged include green leafy and other non-starchy vegetables, nuts, seeds, oils (especially olive oil), fish, poultry, tofu, and avocados. Other foods consistent with the diet include berries (in modest amounts), meats, eggs, and cheese. Key foods to minimize include any sugar-sweetened foods or beverages, bread, pasta, potatoes, highly processed packaged foods, and other starchy foods.
  Interventions: Behavioral: Carbohydrate-restricted diet
- Diet Education + Mindfulness (Experimental): In addition to the carbohydrate-restricted diet described above, the Ed+MBI group will receive mindfulness training consisting of two integrated components: 1) use of a mindful eating app at home to learn and practice mindfulness skills for food-cravings and eating, and 2) in-person group-based meetings to discuss and troubleshoot how the mindfulness practices are working. Key mindfulness content includes helping people improve their relationship with food and control food cravings and using mindful eating approaches including paying attention, noticing habit loops, understanding brain science and food/sugar addiction, disrupting emotional and stress eating, cultivating acceptance and curiosity, lovingkindness, detaching from thoughts, using healthy restraint, and maintaining motivation.
  Interventions: Behavioral: Carbohydrate-restricted diet; Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Carbohydrate-restricted diet — Education for carbohydrate-restricted diet
Behavioral: Mindfulness — Mindful eating app-use and instruction
  Arms: Diet Education + Mindfulness

SUMMARY:
Type 2 diabetes mellitus (T2DM) is the most expensive chronic disease in the U.S.

Lifestyle modification is central to T2DM management, but long-term adherence to dietary recommendations is difficult. A key challenge is the difficulty of coping with cravings for high carbohydrate or sugar-laden foods in an environment where these foods are tempting and widely available. One mechanism by which mindfulness may increase long-term dietary adherence is by better equipping individuals with skills to experience food cravings and difficult emotions without eating in response. Such approaches seek to strengthen abilities to be non-judgmentally aware of, tolerate, and respond skillfully to food cravings and difficult emotions without reacting impulsively or maladaptively. The investigators hypothesize that improved ability to manage food cravings and emotional eating is a key mechanism through which mindfulness-enhancements can improve dietary adherence. The study will test a mindfulness-based intervention (MBI) for improving dietary adherence. Although the particular diet employed is not the focus of this study, the study will use a diet with about 10% of calories from carbohydrate as: (1) it induces a low level of ketone production, which will be used as a biomarker for dietary adherence; (2) prior studies suggest it improves metabolic parameters in T2DM, including glycemic control.

DETAILED DESCRIPTION:
The study will use ecological momentary assessment (EMA) methods to measure eating in response to difficult emotions and/or food cravings. In the R61 phase, the team will ensure this measure is appropriate for further testing and assess the impact of the MBI components on our hypothesized behavioral mechanisms in N=60 persons with T2DM. The study plans 3 waves of 20 persons each with 12 weekly sessions. All participants will attend an in-person group course providing education on basic behavioral strategies for diet and physical activity. Participants will be randomized to receive this education alone (Ed) or this same material with added MBI components (Ed+MBI). The team will also pilot test two levels of intensity of maintenance phase intervention (monthly group meetings alone or supplemented by individualized attention) to prepare them for R33 testing. the investigators plan an R33 phase trial in which 120 persons with T2DM will be randomized (using a 1:2 ratio) to Ed or Ed+MBI conditions and followed for 12 months, including a 9-month maintenance phase. The study will test the robustness of the effect of MBI components on our proposed behavioral mechanisms, and on dietary adherence, as well as preliminary effect sizes on weight and glycemic control. The study will use an innovative adaptive intervention design to optimize maintenance phase intensity, which the investigators believe may be key to augment the MBI effects. The R33 phase will be registered and reported in a separate clinicaltrials.gov record.

ELIGIBILITY:
Inclusion Criteria:

1. History of T2DM mellitus. If taking insulin, screening labs will include C-Peptide to rule out T1DM.
2. HbA1c >= 6.5% and < 12.0% at screening.
3. Experience food-related cravings most days of the week and eat in response to these cravings regularly.
4. Aged 18 years old and older.
5. Able to engage in light physical activity.
6. Willing and able to participate in the interventions. Must be interested in following a carbohydrate- restricted diet, willing to learn about mindful eating and behavioral strategies for following prescribed diets, have sufficient control over their food intake so that they can follow either diet, and otherwise be able and willing to participate in the intervention. Intervention content must be practiced to evaluate whether it is effective.
7. Have smartphone and are willing to use it on a regular basis for data collection.
8. Ability to speak English.

Exclusion Criteria:

1. Unable to provide informed consent.
2. A substance abuse, mental health, or medical condition that, in the opinion of investigators, will make it difficult for the potential participant to participate in the intervention or that may need immediate changes in medical management that will affect study outcome measures. Such conditions may include cancer, liver failure, renal failure, untreated hypo or hyperthyroidism, or history of serious bulimia. Some other serious medical conditions that may alter key study outcomes or require other important diet modifications, including untreated hypothyroidism, renal failure, cirrhosis, and conditions requiring oral or parenteral glucocorticoid treatment.
3. Pregnant or planning to get pregnant in the next 6 months, breastfeeding or less than 6 months post-partum.
4. Current use of weight loss medications, such as Alli or amphetamine-based drugs that may affect weight.
5. Planned weight-loss (bariatric) surgery or bariatric surgery within the past 18 months.
6. Currently enrolled in a weight loss program, such as Weight Watchers or a self-help group such as Overeaters Anonymous, or have unalterable plans to enroll in one of these programs in the next year.
7. Vegan or vegetarian.
8. Unwilling to do home ketone monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rick Hecht, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Osher Center for Integrative Medicine, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mason AE, Saslow LR, Moran PJ, Kim S, Abousleiman H, Richler R, Schleicher S, Goldman VM, Hartman A, Leung C, Hartogensis W, Hecht FM. Lipid findings from the Diabetes Education to Lower Insulin, Sugars, and Hunger (DELISH) Study. Nutr Metab (Lond). 2019 Aug 27;16:58. doi: 10.1186/s12986-019-0383-2. eCollection 2019. PMID 31467583
- [Derived] Mason AE, Saslow L, Moran PJ, Kim S, Wali PK, Abousleiman H, Hartman A, Richler R, Schleicher S, Hartogensis W, Epel ES, Hecht F. Examining the Effects of Mindful Eating Training on Adherence to a Carbohydrate-Restricted Diet in Patients With Type 2 Diabetes (the DELISH Study): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Feb 20;8(2):e11002. doi: 10.2196/11002. PMID 30545813

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment conducted 12/2016-9/2018 via several sources including: flyers posted in and outreach to providers in UCSF clinics (e.g., Diabetes Clinic, General Internal Medicine Clinic); letters mailed to potentially eligible participants in the UCSF system who had previously consented to be contacted about research studies for which they may be eligible; flyers posted in the community as on social media including Facebook, Nextdoor, and Craigslist. First participant was consented 2/17/2017.
Period: Overall Study
Arm/Group | Diet Education | Diet Education + Mindfulness
Started | 28 | 30
Completed | 27 | 28
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diet Education | Diet Education + Mindfulness | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (10.9) | 59.0 (11.2) | 58.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 8 | 13 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Pacific Islander | 7 | 5 | 12
  Black/African-American | 3 | 3 | 6
  Latino/Hispanic | 4 | 2 | 6
  Non-hispanic White | 14 | 15 | 29
  Other/more than 1 race | 0 | 5 | 5
Education [Number; unit: participants]
  High school or less | 1 | 1 | 2
  Some college | 5 | 12 | 17
  4-year college degree | 13 | 7 | 20
  Advanced degree | 9 | 9 | 18
  Declined to report | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Eating in Response to Cravings (Primary Mechanistic Outcome)
Description: Percent of ecological momentary assessment (EMA) opportunities in which participants reported eating in response to food cravings over a 3 day period. EMA measures were delivered to cell phones 3 times each day. The final EMA measure each day included a second question about whether there were any instances of craving related eating not already reported earlier during the day. Thus there was an opportunity to report eating in response to cravings on 4 different EMA questions each day, a total of 12 potential measures over 3 days. The percent here uses the number of EMA responses received as the denominator.
Time Frame: change from baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: % of EMAs with craving related eating
Arm/Group | Diet Education | Diet Education + Mindfulness
Number analyzed (Participants) | 28 | 30
% of EMAs with craving related eating | -20.39 [-28.15 to -12.62] | -25.27 [-32.95 to -17.58]

2. Secondary Outcome: Change in Impulsivity as Measured by Delayed Discounting Score
Description: The 5-trial adaptation of the Delayed Discounting (DD; Koffarnus & Bickel, 2014) is a decision-making exercise where individuals choose between a smaller, immediate reward and a larger, delayed reward. The task measures an individual's "discount rate," or how much they devalue a future reward compared to an immediate one, which is a a key aspect of impulsivity and self-control. Respondents choose between $100 delivered after a delay, or $50 available immediately. To derive estimates of discount rate, we used Mazur's hyperbolic discounting model (V=A/ (1+kD)18, wherein V is the discounted value of the delayed option, A is its objective amount, D is its delay, and k indexes the discount rate. We calculated values of k for each participant as the inverse of the indifference delay (1/ED50). We log transformed these values prior to analysis. Higher values of K indicate greater discounting, which reflects greater impulsivity.
Time Frame: change from baseline to 6 months
Population: Intent to treat; note 2 participants in each arm had impulsivity data excluded due to nonsystematic Delayed Discounting data at baseline
Measure: Geometric Mean (95% Confidence Interval); unit: % change
Arm/Group | Diet Education | Diet Education + Mindfulness
Number analyzed (Participants) | 26 | 28
% change | 87.17 [-38.76 to 472.03] | 6.42 [-63.45 to 209.89]

3. Secondary Outcome: Emotion-related Eating (Secondary Mechanistic Outcome)
Description: Change in emotion-related eating as measured by the Coping subscale of the Palatable Eating Motives Scale (PEMS). The Coping subscale is comprised of 4 items rated on a scale from 1 (almost never/never) to 5 (almost always/always), with possible scores ranging from 4-20. Higher scores reflect worse coping/greater emotional eating. Thus, decreases over time reflect improved coping/decreased emotional eating.
Time Frame: change from baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Diet Education | Diet Education + Mindfulness
Number analyzed (Participants) | 28 | 30
scores on a scale | -0.62 [-1.00 to -0.25] | -0.90 [-1.27 to -0.53]

4. Secondary Outcome: Stress-related Eating (Secondary Mechanistic Outcome)
Description: Change in stress-related eating as measured by two questions about stress-related eating from the MIDUS study. Possible scores range from 2-8. Higher scores reflect worse outcomes/greater eating in response to stress. Thus, decreases over time reflect improved outcomes/decreased stress-related eating.
Time Frame: change from baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Diet Education | Diet Education + Mindfulness
Number analyzed (Participants) | 28 | 30
units on a scale | -1.62 [-2.22 to -1.03] | -1.73 [-2.32 to -1.15]

5. Secondary Outcome: Glycemic Control, Using HbA1c
Description: Change in hemoglobin A1c (HbA1c) from baseline to 6 months by study arm
Time Frame: change from baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: % of hemaglobin with glucose (HbA1C)
Arm/Group | Diet Education | Diet Education + Mindfulness
Number analyzed (Participants) | 28 | 30
% of hemaglobin with glucose (HbA1C) | -1.32 [-1.65 to -0.98] | -0.87 [-1.20 to -0.54]

6. Secondary Outcome: Fasting Glucose
Description: Change in plasma fasting glucose from baseline to 6 months by study arm
Time Frame: change from baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Diet Education | Diet Education + Mindfulness
Number analyzed (Participants) | 28 | 30
mg/dL | -30.21 [-44.48 to -15.94] | -25.92 [-39.67 to -12.17]

7. Secondary Outcome: HOMA-2IR Index of Insulin Resistance (Secondary Clinical Outcome)
Description: Insulin resistance estimated from the Homeostatic model assessment (HOMA) model 2 index of insulin resistance. The basic formula is: (glucose × insulin) / 22.5, where glucose is measured in mmol/L and insulin in mU/L. The computer assisted re-calibration in model 2 addresses variations in the glucose resistance of the peripheral tissue and liver, increases in the insulin secretion curve for glucose > 180 mg/dL, and contribution of circulating pro-insulin. Higher values indicate more insulin resistance (worse outcome). The Oxford University HOMA-2IR calculator was used (https://process.innovation.ox.ac.uk/software/p/2112/homa2-calculator/1). HOMA index values < 2.0 are generally considered normal and indicate adequate sensitivity of cells to insulin. HOMA index values between 2.0 and 2.5 may indicate borderline changes in insulin sensitivity. HOMA index values > 2.5 clearly indicate insulin resistance.
Time Frame: change from baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Diet Education | Diet Education + Mindfulness
Number analyzed (Participants) | 28 | 30
units on a scale | -0.45 [-0.93 to 0.02] | -0.85 [-1.30 to -0.40]

8. Secondary Outcome: Weight Change(Secondary Clinical Outcome)
Description: kilograms
Time Frame: change from baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Diet Education | Diet Education + Mindfulness
Number analyzed (Participants) | 28 | 30
kilograms | -4.96 [-6.44 to -3.49] | -4.43 [-5.88 to -2.98]

9. Secondary Outcome: Adherence to Diet as Measured by Fingerstick Blood Ketones
Description: Adherence to diet as measured by average proportion of fingerstick blood ketones at or above 0.3 mmol/L at 24 weeks.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: proportion of measurements >= 0.3 mmol/L
Arm/Group | Diet Education | Diet Education + Mindfulness
Number analyzed (Participants) | 28 | 30
proportion of measurements >= 0.3 mmol/L | 0.46 [0.26 to 0.66] | 0.60 [0.41 to 0.79]

10. Secondary Outcome: Diet Adherence by Mean Grams of Non-fiber Carbohydrate Consumed Per Day
Description: Diet Adherence Between Intervention Arms as Measured by Mean Grams of Non-fiber Carbohydrate Consumed Per Day From 24- Hour Diet Recall
Time Frame: change from baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: grams
Arm/Group | Diet Education | Diet Education + Mindfulness
Number analyzed (Participants) | 28 | 30
grams | -91.43 [-123.73 to -59.14] | -116.92 [-148.53 to -85.31]

11. Secondary Outcome: Perceived Stress
Description: Perceived Stress Scale (PPS-10) total score. Scores can range from 0 to 40 with higher scores indicated greater perceived stress.
Time Frame: change from baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Diet Education | Diet Education + Mindfulness
Number analyzed (Participants) | 28 | 30
score on a scale | -1.09 [-2.73 to 0.55] | -2.04 [-3.65 to -0.44]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Diet Education | Diet Education + Mindfulness
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/30
Other Adverse Events (participants affected / at risk) | 12/28 | 11/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diet Education (N=28) | Diet Education + Mindfulness (N=30)
Hypoglycemia (Metabolism and nutrition disorders) | 6 (7) | 1 (2)
Hypertriglyceridemia (Cardiac disorders) | 4 (4) | 0 (0)
other (General disorders) | 6 (9) | 11 (14)

LIMITATIONS AND CAVEATS:
We completed planned enrollment and did not have early termination. The trial was the initial part of a potentially two-step grant. This pilot phase was aimed at testing the trial design and assessing if there was evidence of effects on food cravings, a mechanistic goal. It was not powered to assess changes in clinical outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/11/NCT03207711/Prot_SAP_001.pdf
  • Informed Consent Form (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT03207711/ICF_002.pdf